CLINICAL TRIAL: NCT05848882
Title: Comparison Between Removable Devices in Palatal Expansion: a Randomized Open Label Clinical Trial
Brief Title: Removable Devices in Palatal Expansion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Eleonora Ortu, Principal Investigator, University of L'Aquila
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB L'Aquila 57/2021-2022
Record Dates: First submitted 2023-04-27; First posted 2023-05-08 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Palatal Expansion Technique
Keywords: elastodontic device; growing patients; transversal palatal discrepancies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elastodontic removable device (Experimental): Patients in this group will be treat with an elastodontic device adapted to the patient according to the shape of the dental arches. This device is similar to a mouthguard and embraces both dental arches. This appliance is worn overnight and the patient will be checked every month. The distance between the palatal cusps of the first upper premolars will be taken at T0( before the start of the therapy), at T1 (after six months)and at T2 (after one month). All the dental recors will be taken by the same operator with an intraoral scanner 3D.
  Interventions: Device: Elastodontic Device
- Schwarz removable device (Experimental): Patients in this group will be treat with a Schwarz removable device constructed individually by the dental technician.This device has a resin baseplate with an activation screw in the center and Adams hooks on the upper first molars and it works by turning the expansion screw in the center of the palate one-quarter turn, once or twice a month by the ortodontist. This appliance is worn overnight and some hours during the day (totally 16 hours).The distance between the palatal cusps of the first upper premolars will be taken at T0( before the start of the therapy), at T1 (after six months)and at T2 (after one month). All the dental recors will be taken by the same operator with an intraoral scanner 3D.
  Interventions: Device: Elastodontic Device

INTERVENTIONS:
Device: Elastodontic Device — Removable device that embraces two dental archs

SUMMARY:
The goal of this clinical trial si to compare two removable devices used to treat the transversal discrepancies in growing patients.

The main questions it aims to answer are:

* the efficacy of the two devices in the palatal expansion
* the neuromuscolar effects developed on the stomatognatic system Participants will be instructed in the use and maintenance of the devices and will be checked every 15-30 days for one year.

ELIGIBILITY:
Inclusion Criteria:

skeletal class I relationship, molar class I relationship; complete eruption of upper first premolars ; presence of unilateral or bilateral cross bite (falling within grade 3 IOTN index)

Exclusion Criteria:

IOTN index >4; presence of temporomandibular disorders, epilepsy, systemic diseases, periodontal disease, absence of written informed consent signed by parents/legal guardians

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Palatal first premolars width | 12 months
  To compare the palatal first premolars width in three times

CONTACTS AND LOCATIONS:
Locations (1):
- Dipartimento MeSVA, L’Aquila, Aq, Italy

IPD SHARING:
Plan to Share IPD: No